CLINICAL TRIAL: NCT00177385
Title: AGEWISE Project 4: PROTECTING HEALTH IN LATER LIFE
Brief Title: Aging Well, Sleeping Efficiently: Protecting Health In Later Life
Acronym: AgeWise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #021116; 5P01AG020677 (NIH); 5P01AG020677-05 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Sleep; Health Promotion
Keywords: Sleep; Sleep Hygiene; Modest sleep deprivation; Healthy Aging and sleep; Health Promotion
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Modest sleep deprivation with sleep hygiene education

SUMMARY:
The purpose of this study is to see whether protecting sleep quality in later life is important in continued healthy aging. The value of education in healthy sleep practices along with reducing time in bed each night by going to bed 30 minutes later, and of healthy dietary practices will be tested for their effects on sleep quality, health, and well being.

DETAILED DESCRIPTION:
The goal of this project is to test the efficacy of restricting time in bed and education in healthy sleep practices for maintaining or even enhancing sleep consolidation and depth in subjects aged 75+ who are at risk for decay in sleep quality and daytime well being; to determine the associated benefits for health; and to examine the persistence of such effects for 12 months beyond the end of the 18-month intervention. This project focuses not on pathology but on prevention of sleep decay and preservation of sleep in individuals who have already evidenced successful aging.

ELIGIBILITY:
Inclusion Criteria:

* age 75 or older
* without sleep disorders
* without psychiatric disorders
* Folstein MMSE of 24 or greater

Exclusion Criteria:

* Apnea-hypopnea index greater than 30
* Mean sleep latency less than 6
* Psychotropic medications present

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66
Dates: Start 2003-06; Primary Completion 2009-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Polysomnographic measures of sleep consolidation, sleep depth and daytime sleepiness at baseline, 6mos.,12mos., 18mos.,30 mons.

SECONDARY OUTCOMES:
Clinical measures of sleep quality, general functioning, mental health at baseline,6 mos., 12 mons., 18mons.,30mons.

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. Reynolds lll, M.D., Principal Investigator — University of Pittsburgh Medical Center

REFERENCES:
- See also: AgeWise Program Description — http://www.aging.upmc.com/aging-well.htm